CLINICAL TRIAL: NCT03236662
Title: UCD0115B: An Open-label Extension Study of Purified Epicatechin to Improve Mitochondrial Function, Strength and Skeletal Muscle Exercise Response in Becker Muscular Dystrophy
Brief Title: (-)- Epicatechin Becker Muscular Dystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Craig McDonald, MD (Other)
Collaborators: Cardero Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Craig McDonald, MD, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 767161
Record Dates: First submitted 2016-11-07; First posted 2017-08-02 (Actual); Results first posted 2021-07-26 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Becker Muscular Dystrophy
Keywords: BMD; Becker muscular dystrophy; epicatechin; clinical trial; neuromuscular disease
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Neuromuscular Diseases | interventions — Catechin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): (-)-epicatechin 50mg twice per day (100mg per day total dose)
  Interventions: Drug: (-)-Epicatechin

INTERVENTIONS:
Drug: (-)-Epicatechin

SUMMARY:
This is a 48-week open-label extension of our initial proof-of-concept study (UCD0113) in patients with Becker muscular dystrophy who participated in the earlier trial. This single center study will enroll up to 10 adults who will receive the purified nutritional extract (-)-epicatechin 100mg/day orally for 8 weeks. After screening visits, participants will be enrolled in the study if they meet all inclusion criteria. They will be evaluated at screening, baseline, and weeks 4, 8, 12, 24, 16 and 48. The main criterion for success of the study will be presence of one or more biologic or strength and performance outcome measures that yield a response magnitude that allows for sufficient power in a Phase II B study with a sample size of 30 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Prior participation in UCD0113 BMD epicatechin pilot study
* Male
* Age 18 years to 70 years
* Average to low daily physical activity
* Ability to ambulate for 75 meters without assistive devices
* Diagnosis of BMD confirmed by at least one the following:
* Dystrophin immunofluorescence and/or immunoblot showing partial dystrophin deficiency, and clinical picture consistent with typical BMD, or
* Gene deletions test positive (missing one or more exons) of the dystrophin gene, where reading frame can be predicted as 'in-frame', and clinical picture consistent with typical BMD, or
* Complete dystrophin gene sequencing showing an alteration (point mutation, duplication, or other mutation resulting in a stop codon mutation) that can be definitely associated with BMD, with a typical clinical picture of BMD, or
* Positive family history of BMD confirmed by one of the criteria listed above in a sibling or maternal uncle, and clinical picture typical of BMD.
* Hematology profile within normal range
* Baseline laboratory safety chemistry profile within normal range
* No plan to change exercise regimen during study participation
* Nutritional, herbal and antioxidant supplements taken with the intent of maintaining or improving skeletal muscle strength or functional mobility have been discontinued at least 2 weeks prior to screening (daily multivitamin use is acceptable).

Exclusion Criteria:

* Currently enrolled in another treatment clinical trial.
* History of significant concomitant illness or significant impairment of renal or hepatic function.
* Use of regular daily aspirin or other medication with antiplatelet effects within 3 weeks of first dose of study medication.
* Regular participation in vigorous exercise.
* Symptomatic heart failure with cardiac ejection fraction <25%

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: (-)-epicatechin 50mg twice per day (100mg per day total dose)
  (-)-Epicatechin
Period: Overall Study
Arm/Group | Treatment
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 54 [52 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Plasma Follistatin
Description: blood biomarker concentration
Time Frame: 48 weeks
Population: Due to lack of funding, only 2 participants could be enrolled. The number of evaluable patients was insufficient to perform analysis of this outcome measure.
Arm/Group | Treatment
Number analyzed (Participants) | 0

2. Primary Outcome: Plasma Myostatin
Description: blood biomarker concentration
Time Frame: 48 weeks
Population: as for outcome 1
Arm/Group | Treatment
Number analyzed (Participants) | 0

3. Primary Outcome: Plasma Nitrates/ SNO
Description: blood biomarker concentration
Time Frame: 48 weeks
Population: as for outcome 1
Arm/Group | Treatment
Number analyzed (Participants) | 0

4. Primary Outcome: Plasma BNP
Description: blood biomarker concentration
Time Frame: 48 weeks
Population: as for outcome 1
Arm/Group | Treatment
Number analyzed (Participants) | 0

5. Primary Outcome: Plasma Creatine Kinase
Description: blood biomarker concentration
Time Frame: 48 weeks
Population: as for outcome 1
Arm/Group | Treatment
Number analyzed (Participants) | 0

6. Primary Outcome: Plasma MMP-9
Description: blood biomarker concentration
Time Frame: 48 weeks
Population: as for outcome 1
Arm/Group | Treatment
Number analyzed (Participants) | 0

7. Primary Outcome: Plasma TNF-Alpha
Description: blood biomarker concentration
Time Frame: 48 weeks
Population: as for outcome 1
Arm/Group | Treatment
Number analyzed (Participants) | 0

8. Primary Outcome: Plasma TGF-Beta
Description: blood biomarker concentration
Time Frame: 48 weeks
Population: as for outcome 1
Arm/Group | Treatment
Number analyzed (Participants) | 0

9. Primary Outcome: Plasma Follistatin:Myostain Ratio
Description: Ratio of plasma follistatin to plasma myostatin
Time Frame: 48 weeks
Population: as for outcome 1
Arm/Group | Treatment
Number analyzed (Participants) | 0

10. Secondary Outcome: Graded Exercise Test Using a Recumbent Cycle Ergometer
Description: blood lactate measured
Time Frame: baseline and at 2-minute intervals
Population: as for outcome 1
Arm/Group | Treatment
Number analyzed (Participants) | 0

11. Secondary Outcome: 6-minute Walk Test
Description: Measurements recorded will include 25-meter split times and total distance traveled.
Time Frame: 48 weeks
Population: as for outcome 1
Arm/Group | Treatment
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Exploratory Proteomics
Description: Collection of plasma samples for proteomics analysis.
Time Frame: 48 weeks
Population: as for outcome 1
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-06-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT03236662/Prot_SAP_002.pdf
  • Informed Consent Form (2015-08-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT03236662/ICF_001.pdf